CLINICAL TRIAL: NCT04533477
Title: Application and Efficacy of Reconstructing Forked Corpus Spongiosum in Hypospadias Repair
Brief Title: Reconstructing Forked Corpus Spongiosum in Hypospadias Repair
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Principal Investigator, Zhangbin, Principal Investigator, Children's Hospital of Fudan University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Zhangbin_001
Record Dates: First submitted 2020-08-24; First posted 2020-08-31 (Actual); Last update posted 2022-08-10 (Actual); Status verified 2022-08

CONDITIONS: Hypospadias
Keywords: Hypospadias repair; Forked corpus spongiosum
MeSH Terms: conditions — Hypospadias

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Routine surgery with reconstructing FCS (Experimental): The participants undergo FCS reconstruction during the routine standardized surgery.
  Interventions: Procedure: Reconstructing forked corpus spongiosum (FCS); Procedure: Routine standardized surgery
- Routine surgery (Active Comparator): The participants undergo routine standardized surgery.
  Interventions: Procedure: Routine standardized surgery

INTERVENTIONS:
Procedure: Reconstructing forked corpus spongiosum (FCS) — During the routine standardized surgery, the FCS should be cut off along both sides of the middle urethral plate before dissecting the glans wings and then dissected along the penile tunica albuginea closely from the near to the far side of the penis until the top of the penis head was reached. The corpus spongiosum on both sides will be reserved for the two wings of the glans. The two wings of the glans should be carefully expanded to at least the 3 o'clock and 9 o'clock positions of the penis. Some cases of small glans should be dissected to the 2 o'clock and 10 o'clock positions to close the two wings of the glans with no tension when performing glansplasty. Additionally, the original FCS on both sides should be combined at the coronal sulcus, thereby covering the surface of the new urethra.
  Arms: Routine surgery with reconstructing FCS
Procedure: Routine standardized surgery — When the urethral plate can be preserved after degloving, the investigators chose the surgical method according to the width of the urethral plate. If the width of the urethral plate is ≥6 mm, tubularized incised plate (TIP) urethroplasty will be performed, whereas if the width of the urethral plate is <6 mm, the onlay island flap (ONLAY) technique will be performed. When the urethral plate can not be preserved after degloving, transverse preputial island flap urethroplasty (Duckett) will be performed.

SUMMARY:
Hypospadias is one of the most common genital malformations in children. The high incidence of hypospadias, which occurs in 1 in 200 to 300 live births, means that it affects a large number of patients. Surgery is the only way to repair hypospadias. Over 400 techniques have been described for hypospadias repair. However, the surgical success rate of hypospadias is still not ideal. Although the surgical success rate of distal hypospadias has reached more than 85%, the complications of proximal hypospadias are still as high as 30-68%. How to improve surgical skills and reduce the postoperative complications is quite a challenge for pediatric urologists.

In the preliminary clinical work, the investigators have tried to apply the technique of reconstructing forked corpus spongiosum (FCS) in hypospadias repair with urethral plate preservation. It has been confirmed that this technique was effective in reducing postoperative complications of this type of hypospadias repair. In order to promote the technology of reconstructing FCS, the investigators need to perform this technology in various types of hypospadias and evaluate its true effectiveness. Therefore, the investigators need to design a prospective, randomized, parallel-controlled, single-blind, and superior clinical trial to analyze the efficacy of reconstructing FCS in hypospadias repair.

In this study, the investigators will perform one-stage surgical repair on children with primary hypospadias by the same surgeon in Urology Department, Children's Hospital of Fudan University, Shanghai, China. Participants will be random grouped: Routine standardized surgery with reconstructing FCS group and Routine standardized surgery group. All participants will be closely followed up and regularly evaluated after surgery, including postoperative complications, HOSE objective score of cosmetic outcome and voiding function. By collecting all data and conducting statistical analysis, the investigators will evaluate the followings: (1) the correlation between the penile curvature and the development of FCS; (2) the effect of reconstructing FCS on the complications of primary hypospadias repair; (3) the effect of reconstructing FCS on the cosmetic outcome; (4) the influence of reconstructing FCS on postoperative voiding function.

Based on this clinical randomized controlled study, the investigators intend to prove the feasibility and effectiveness of the new technology of reconstructing FCS in various types of hypospadias repair. The study will provide a reliable basis for the promotion of this technology for hypospadias repair in order to improve the quality of life for children with hypospadias.

ELIGIBILITY:
Inclusion Criteria:

* children with primary hypospadias
* one-stage surgical repair

Exclusion Criteria:

* staged surgery repair
* micropenis
* reoperation for postoperative complications
* using testosterone or male hormones preoperatively

Ages: 6 Months to 15 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 260 (Estimated)
Dates: Start 2023-03-01 (Estimated); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Postoperative complications | 1 to 6 months after surgery
  It is a binary variable (1/0) that needs repeated measurement. The variable would be setted into "1", if any complications including residual chordee, fistula, diverticulum, glans dehiscence, meatus stenosis, or urethral stricture happeded.

SECONDARY OUTCOMES:
Residual chordee | 1 to 6 months after surgery
  It is a binary variable (1/0) that needs repeated measurement. The variable would be setted into "1", if residual chordee happeded.
Fistula | 1 to 6 months after surgery
  It is a binary variable (1/0) that needs repeated measurement. The variable would be setted into "1", if fistula happeded.
Diverticulum | 1 to 6 months after surgery
  It is a binary variable (1/0) that needs repeated measurement. The variable would be setted into "1", if diverticulum happeded.
Glans dehiscence | 1 to 6 months after surgery
  It is a binary variable (1/0) that needs repeated measurement. The variable would be setted into "1", if glans dehiscence happeded.
Meatus stenosis | 1 to 6 months after surgery
  It is a binary variable (1/0) that needs repeated measurement. The variable would be setted into "1", if meatus stenosis happeded.
Urethral stricture | 1 to 6 months after surgery
  It is a binary variable (1/0) that needs repeated measurement. The variable would be setted into "1", if urethral stricture happeded.
Hypospadias objective scoring evaluation | at 6 month after surgery
  It is an objective scoring system for evaluating the cosmetic outcome of hypospadias surgery. The scoring system is designed so that the minimum total score would be 5, corresponding to a worst score for each variable, to a maximum total of 16, equivalent to the best score for each variable.

IPD SHARING:
Plan to Share IPD: No